CLINICAL TRIAL: NCT06231823
Title: The Extraction of Compromised First Permanent Molars in a Group of Egyptian Children
Brief Title: Extraction of the Compromised First Permanent Molars
Acronym: FPM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dina darwish, lecturer, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDASU-RecIR012364
Record Dates: First submitted 2024-01-15; First posted 2024-01-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Caries; Caries,Dental
Keywords: first permanent molar; molar incisor hypo mineralization; dental extraction; space closure
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- extraction of the compromised first permanent molars at 8-10 years children (Experimental): extraction of badly decayed FPM at the E,F developmental stages of the second permanent molar.
  Interventions: Other: Extraction

INTERVENTIONS:
Other: Extraction — Simple / surgical dental extraction for necrotic. irreversible pulpitis, unrestorable, and first permanent molars with sever molar incisor hypomineralization.

SUMMARY:
Compromised first permanent molars (FPM), whether diagnosed with severe molar incisor hypomineralization (MIH), irreversible pulpities, or necrosis, require frequent re-treatment consequently entering the restorative cycle, which leads to their inevitable extraction and implant placement. Extraction of compromised first permanent molars in 8-10-year-old children allows the mesial migration of the second permanent molars during their eruption, thereby favoring spontaneous space closure as a permanent solution.

DETAILED DESCRIPTION:
Extraction of compromised first permanent molars in children decreases the burden of repeated restorative procedures for theses molars, which will eventually need frequent repair. This will end in their inevitable extraction with its consequences. The extraction of the FPM will be delivered by Nour Wahba, Dina Darwish, and Basma Nagi, lecturers in Pediatric Dentistry and Dental Public Health Department, faculty of Dentistry, Ain Shams University.All patients will be recalled for follow-up yearly for three-years. The first follow-up will be done after 6months to perform the Quality of life questionnaires. The position of the second permanent molar will be checked clinically and radiographically to evaluate the space between second premolar and the second molar.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients' class I according to the American Society of Anesthesiologists (ASA class I)
* Age: 8-10 years
* Angle class I occlusion
* The radiographic presence of the second premolar
* The radiographic stages of development E or F for formation the second permanent molar.
* First permanent molar that is severely affected by MIH, signs of necrosis, signs of irreversible pulpitis or non-restorability.

Exclusion Criteria:

* Refusal of the parents to sign the informed consent.
* Signs of reversible pulpitis of first permanent molar.
* Patients with severe malocclusion.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 37 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
clinical spontaneous space closure | 3 years
  Clinically, using periodontal probe measure the amount of space between the distal surface of second premolar and mesial surface of second permanent molar.
radiographic spontaneous space closure | 3 years
  radiographically, using panoramic radiograph

SECONDARY OUTCOMES:
assessment of the Quality of life | 6 months
  Measure the quality of life of the children before extraction and at 6 months follow-up using parent perception questionnaire and family impact scale (P-CPQ and FIS) and child perception questionnaire 8- 10 or 11-14 (CPQ 8-10; CPQ 11-14) according to the child's age.
Midline shift | 3 years
  Investigate the midline shift by clinical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Dina D Abdelmoneim, Principal Investigator — Ain Shams Univeristy
Locations (1):
- Ain Shams University, Cairo, El-Willi, Egypt

IPD SHARING:
Plan to Share IPD: No